CLINICAL TRIAL: NCT04602052
Title: Comparison of Surgical Versus Medical Termination of Pregnancy Between 13-20 Weeks of Gestation in Ethiopia: A Quasi-experimental Study.
Brief Title: Comparison of Surgical Versus Medical Termination of Pregnancy Between 13-20 Weeks of Gestation in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital Millennium Medical College, Ethiopia (Other)
Responsible Party: Principal Investigator, Tesfaye H. Tufa, MD, Assistant Professor of Obstetrics and Gynecology, St. Paul's Hospital Millennium Medical College, Ethiopia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StPaulsHMM
Record Dates: First submitted 2020-10-14; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Termination of Pregnancy
Keywords: Dilation and evacuation; Second Trimester; Medical abortion; Ethiopia
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Dilatation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical arm (Active Comparator): Those who choose medical abortion receive mifepristone 200 mg on day 1 and are appointed to return to SPHMMC 24-48 hours later for admission and misoprostol administration.
  Interventions: Procedure: Dilation and evacuation
- Surgical arm (Experimental): Those who chose surgical abortion are given mifepristone 200 mg with or without laminaria and appointed to return the next day for surgical abortion.
  Interventions: Procedure: Dilation and evacuation

INTERVENTIONS:
Procedure: Dilation and evacuation — Abortion is termination of pregannacy by evaccuating the uterus using either medical or surgical technique
  Other Names: Medical abortion

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of dilation and evacuation for surgical abortion as compared to medical abortion

DETAILED DESCRIPTION:
All patients with a gestational age between 13-20 weeks are fully counseled on the risks and benefits and given the option of medical or surgical abortion. Those who choose medical abortion receive mifepristone 200 mg on day 1 and are appointed to return to SPHMMC 24-48 hours later for admission and misoprostol administration. Those who chose surgical abortion are given mifepristone 200 mg with or without laminaria and appointed to return the next day for surgical abortion.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 13 - 20 weeks confirmed with ultrasound,
* Age at or more than18 years,
* Having a working phone and willingness to be contacted for a follow-up questionnaire 2 weeks after the procedure.

Exclusion criteria

* Inability to give consent
* complicated abortion (missed abortion, septic abortion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Composite complication rate | During the abortion procedure and within 2 weeks post procedure
  Presence of one of the following complications: bleeding requiring observation, genital tract lacerations requiring repair, need for additional intervention to complete the abortion procedure, and one or more symptoms of pelvic infection

SECONDARY OUTCOMES:
Other serious maternal complications | During the abortion procedure and within 2 weeks post procedure
  Continued bleeding for more than two weeks, additional major surgery (laparotomy), and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Information can be shared up on request
Supporting Information: CSR
Time Frame: Currently available